CLINICAL TRIAL: NCT06073054
Title: A Pharmacist Intervention to Improve Mother and Child Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Hao P. Tran, Clinical Assistant Professor, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 202305322; 1UM1TR004403-01 (NIH)
Record Dates: First submitted 2023-09-22; First posted 2023-10-10 (Actual); Results first posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Research Pharmacist Monitoring (Experimental): The pharmacist will help the mother find a primary care physician if she doesn't have one, obtain health insurance if she doesn't have any, and discuss any health-related information about herself or her child, as needed. These pharmacist interactions will occur 7 days after baseline and again 1 month later (the participant will be asked to measure and text their blood pressure again 1 time per day for 3 days during the follow-up month). If the participant's blood pressures become elevated, the pharmacist will provide behavioral and lifestyle interventions to attempt to lower the blood pressure. They may also recommend medications to the participant's physician. The pharmacist will have access to the participant's electronic medical record to obtain any blood pressure-related medications that the mother is prescribed as well as throughout the follow up to ensure any health-related conditions can be discussed, as necessary.
  Interventions: Behavioral: Research Pharmacist

INTERVENTIONS:
Behavioral: Research Pharmacist — The goal of this intervention is to determine if contact with the research pharmacist will improve the health of the mother and/or child.

SUMMARY:
The goal of this clinical trial is to learn if a research pharmacist can improve the health of new mothers and their babies. The main questions it aims to answer are:

* Will postpartum women who had elevated blood pressure during pregnancy be willing to participate in the study, talk to a pharmacist about their health and the health of their child, and text us their blood pressure measurements?
* Will contact with the pharmacist improve the health of the mother and/or the child?

Participants will:

* complete a baseline demographic survey,
* be given a blood pressure cuff and taught how to use it,
* be asked to text us their blood pressure values 2 times per day for 7 days after enrollment,
* complete a phone call with a pharmacist discussing their health and the health of their baby,
* text us their blood pressure 1 time per day for 3 days 1 month after enrollment,
* have a 1 month follow-up phone call with the research pharmacist, and
* complete an exit survey to provide feedback about the study.

ELIGIBILITY:
Inclusion Criteria:

* biological mother of a baby attending a 1-week to 6-month well-child visit,
* received prenatal care at University of Iowa Hospitals and Clinics,
* had at least 2 elevated blood pressures (>= 130 mmHg systolic or >= 80 mmHg diastolic) during pregnancy,
* owns a smartphone

Exclusion Criteria:

* arm circumference > 17 inches,
* prisoner status
* unable to provide own written informed consent

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 25 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hao Tran, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Research Pharmacist Monitoring
Started | 25
Completed | 23
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Research Pharmacist Monitoring
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 17
  More than one race | 0
  Unknown or Not Reported | 2
Education [Count of Participants; unit: Participants]
  High School | 1
  Some College/Associate's | 5
  Bachelor's | 11
  Master's | 6
  Doctoral Degree | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Talk to Research Pharmacist
Description: We will calculate the number of participants who talk to the research pharmacist during the course of the intervention.
Time Frame: Through study completion, an average of 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Research Pharmacist Monitoring
Number analyzed (Participants) | 25
Participants | 20

2. Primary Outcome: Number of Participants Who Return BP Measurements
Description: We will calculate the number of participants who return at least one blood pressure measurement via text message.
Time Frame: Through study completion, an average of 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Research Pharmacist Monitoring
Number analyzed (Participants) | 25
Participants | 22

3. Primary Outcome: Percentage of Well-Child Visits Attended
Description: We will calculate the percentage of well-child visits that are attended by each family.
Time Frame: Through study completion, an average of 30 days
Measure: Count of Units; unit: Well-child visits
Units Other Than Participants: Well-child visits
Arm/Group | Research Pharmacist Monitoring
Number analyzed (Participants) | 25
Number analyzed (Well-child visits) | 65
Well-child visits | 57

4. Primary Outcome: Percentage of Vaccinations Received
Description: We will calculate the percentage of vaccinations received by each child.
Time Frame: Through study completion, an average of 30 days
Measure: Count of Units; unit: Vaccinations
Units Other Than Participants: Vaccinations
Arm/Group | Research Pharmacist Monitoring
Number analyzed (Participants) | 25
Number analyzed (Vaccinations) | 300
Vaccinations | 251

5. Secondary Outcome: Number of BP Measurements Submitted
Description: We will calculate the number of blood pressure values that are submitted by each participant.
Time Frame: Through study completion, an average of 30 days
Measure: Mean (Standard Deviation); unit: Mean Number of Blood Pressure Values
Arm/Group | Research Pharmacist Monitoring
Number analyzed (Participants) | 23
Mean Number of Blood Pressure Values | 12.9 (5.3)

6. Secondary Outcome: Blood Pressure Control
Description: We will determine how many participants' blood pressure is controlled after the intervention.
Time Frame: Through study completion, an average of 30 days
Population: Only 13 participants provided information on blood pressure control at the end of the study, but they did not withdraw from the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Research Pharmacist Monitoring
Number analyzed (Participants) | 13
Participants | 12

7. Secondary Outcome: Number of Participants Satisfied With the Study
Description: We will measure participant satisfaction with the study using an exit survey. Satisfaction will be measured by a response of Extremely Helpful or Helpful on the question- My contact(s) with the pharmacist about my health were....
Time Frame: Through study completion, an average of 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Research Pharmacist Monitoring
Number analyzed (Participants) | 11
Participants | 7

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Research Pharmacist Monitoring
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT06073054/Prot_SAP_000.pdf
  • Informed Consent Form (2025-07-23): https://cdn.clinicaltrials.gov/large-docs/54/NCT06073054/ICF_001.pdf